CLINICAL TRIAL: NCT00270699
Title: Phase 1 Study of the Safety and Immunogenicity of rDEN4delta30-200,201, a Live Attenuated Virus Vaccine Candidate for the Prevention of Dengue Serotype 4
Brief Title: Safety of and Immune Response to a Dengue Virus Vaccine (rDEN4delta30-200,201) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 214; WIRB Protocol Number 2006478
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Dengue Fever
Keywords: Dengue Vaccine; Dengue Virus; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): One subcutaneous vaccination with rDEN4delta30-200,201 vaccine (10^5 PFU dose) into the deltoid region of either arm.
  Interventions: Biological: rDEN4delta30-200,201
- 2 (Experimental): One subcutaneous vaccination with rDEN4delta30-200,201 vaccine (10^3 PFU dose) into the deltoid region of either arm. This arm will enroll after Arm 1.
  Interventions: Biological: rDEN4delta30-200,201
- 3 (Experimental): One subcutaneous vaccination with rDEN4delta30-200,201 vaccine (10^1 PFU dose) into the deltoid region of either arm. This arm will enroll after Arms 1 and 2.
  Interventions: Biological: rDEN4delta30-200,201
- 4 (Placebo Comparator): One subcutaneous vaccination with placebo into the deltoid region of either arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rDEN4delta30-200,201 — Live attenuated dengue 4 vaccine (one of three doses)
  Arms: 1; 2; 3
Biological: Placebo — Placebo for rDEN4delta30-200,201
  Arms: 4

SUMMARY:
Dengue fever, which is caused by dengue viruses, is a major health problem in tropical and subtropical regions of the world. The purpose of this study is to test the safety of and immune response to a new dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses cause dengue fever and the more severe dengue hemorrhagic fever/shock syndrome. More than 2 billion people living in tropical and subtropical regions of the world are at risk of dengue virus infection, which is the leading cause of hospitalization and death in children in several tropical Asian countries. This study will evaluate the safety and immunogenicity of a live attenuated dengue virus vaccine called rDEN4delta30-200,201. This vaccine is derived from rDEN4delta30, another dengue virus vaccine candidate that has been shown to be safe and immunogenic in Phase I and II trials in healthy adults.

This study will last 180 days. There will be three cohorts in this dose de-escalation study. Participants in Cohort 1 will be randomly assigned to receive the highest dose of rDEN4delta30-200,201 or placebo at study entry. Cohort 2 will begin only after safety review of all participants in Cohort 1. Participants in Cohort 2 will receive a lower dose of rDEN4delta30-200,201 or placebo. Cohort 3 will begin only after safety review of all participants in Cohort 2. Participants in Cohort 3 will receive the lowest dose of rDEN4delta30-200,201 or placebo.

After vaccination, participants will be asked to monitor their temperatures every day for 16 days. Study visits will occur every other day after vaccination until Day 16, followed by four additional visits at selected days through Day 180. Blood collection, vital signs measurement, and a targeted physical exam will occur at each study visit. Some participants will be asked to undergo a skin biopsy or additional blood collection at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be followed for the duration of the study
* Willing to use acceptable methods of contraception
* Good general health

Exclusion Criteria:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, may affect the ability of the volunteer to understand and cooperate with the study
* Laboratory abnormalities at study screening
* Alcohol or drug abuse within 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Emergency room visit or hospitalization for severe asthma within 6 months prior to study entry
* HIV-1 infected
* Hepatitis C virus infected
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days prior to study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Blood products within 6 months prior to study entry
* Previously received a licensed or experimental yellow fever or dengue vaccine
* Surgical removal of spleen
* History of dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, West Nile virus, Japanese encephalitis virus)
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study
* Plan to travel to an area where dengue infection is common
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse events, as classified by intensity and severity through active and passive surveillance and separate assessments of systemic and local reactions | Throughout study
Determine the number of vaccinees who have seroconverted to DEN4 up to and including Day 42 | At 42 days

SECONDARY OUTCOMES:
Durability of antibody responses to DEN4 virus | At 180 days
Frequency, quantity, and duration of viremia in each dose cohort | Thoughout study
Number of vaccinees infected with vaccine virus in each dose cohort | Throughout study
Duration of antibody response determined by serum neutralizing antibody | At 180 days
Determine cellular targets of vaccine infection in participants willing to undergo skin biopsy | Throughout study
Compare infectivity rates, safety, and immunogenicity between dose cohorts | At study completion
Evaluate immunopathological mechanism of vaccine-associated rash in participants willing to undergo skin biopsy | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, Johns Hopkins School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Durbin AP, Whitehead SS, McArthur J, Perreault JR, Blaney JE Jr, Thumar B, Murphy BR, Karron RA. rDEN4delta30, a live attenuated dengue virus type 4 vaccine candidate, is safe, immunogenic, and highly infectious in healthy adult volunteers. J Infect Dis. 2005 Mar 1;191(5):710-8. doi: 10.1086/427780. Epub 2005 Jan 27. PMID 15688284
- [Background] Guzman MG, Mune M, Kouri G. Dengue vaccine: priorities and progress. Expert Rev Anti Infect Ther. 2004 Dec;2(6):895-911. doi: 10.1586/14789072.2.6.895. PMID 15566333
- [Background] Malavige GN, Fernando S, Fernando DJ, Seneviratne SL. Dengue viral infections. Postgrad Med J. 2004 Oct;80(948):588-601. doi: 10.1136/pgmj.2004.019638. PMID 15466994
- [Background] Rothman AL. Dengue: defining protective versus pathologic immunity. J Clin Invest. 2004 Apr;113(7):946-51. doi: 10.1172/JCI21512. PMID 15057297
- [Background] Sun W, Edelman R, Kanesa-Thasan N, Eckels KH, Putnak JR, King AD, Houng HS, Tang D, Scherer JM, Hoke CH Jr, Innis BL. Vaccination of human volunteers with monovalent and tetravalent live-attenuated dengue vaccine candidates. Am J Trop Med Hyg. 2003 Dec;69(6 Suppl):24-31. doi: 10.4269/ajtmh.2003.69.6_suppl.0690024. PMID 14740952